CLINICAL TRIAL: NCT03912831
Title: A Phase 1 Study Evaluating the Safety and Efficacy of HPV16 E7 T Cell Receptor Engineered T Cells (KITE-439) in HLA-A*02:01+ Subjects With Relapsed/Refractory HPV16+ Cancers
Brief Title: Study to Evaluate the Safety and Efficacy of KITE-439 in HLA-A*02:01+ Adults With Relapsed/Refractory HPV16+ Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program terminated
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-478-0401
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Human Papillomavirus (HPV) 16+ Relapsed/Refractory Cancer
MeSH Terms: conditions — Papillomavirus Infections; Neoplasms | interventions — Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) (Experimental): Participants will receive conditioning chemotherapy of cyclophosphamide 30 mg/kg, intravenous (IV) infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^6 E7 T-cell receptor (TCR) T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, subcutaneous (SC) injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) (Experimental): Participants will receive conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 3 × 10^6 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) (Experimental): Participants will receive conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^7 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) (Experimental): Participants will receive conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 3 × 10^7 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) (Experimental): Participants will receive conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^8 E7 TCR T cells/kg on Day 0 (maximum allowable dose is 5 × 10^9 E7 TCR T cells) along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Phase 1A: 1 x 10^8 KITE-439 (Cohort 6) (Experimental): Participants will receive conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^8 E7 TCR T cells/kg on Day 0 (maximum allowable dose is 1 × 10^10 E7 TCR T cells) along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2
- Phase 1B: KITE-439 (Experimental): Participants will receive cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, at a dose selected based on Phase 1A along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
  Interventions: Drug: KITE-439; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2

INTERVENTIONS:
Drug: KITE-439 — A single infusion of E7 TCR T cells (KITE-439).
Drug: Cyclophosphamide — Administered intravenously.
Drug: Fludarabine — Administered intravenously.
Drug: Interleukin-2 — Administered subcutaneously.

SUMMARY:
This study has 2 parts: Phase 1A and Phase 1B. The primary objectives of Phase 1A are to evaluate the safety of KITE-439 and to determine a recommended Phase 1B dose. The primary objective of Phase 1B is to estimate the efficacy of KITE-439 in adults who are human leukocyte antigen (HLA)-A*02:01+ and have relapsed/refractory human papillomavirus (HPV)16+ cancers.

ELIGIBILITY:
Key Inclusion Criteria:

* Advanced cancer defined as relapsed or refractory disease after at least 1 line of therapy that included systemic chemotherapy and that is not amenable to definitive locoregional therapy
* HPV16+ tumor as confirmed by the central laboratory
* HLA type is HLA-A*02:01+ per local assessment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Key Exclusion Criteria:

* Presence of fungal, bacterial, viral, or other infection requiring anti-microbials for management

  * Note: Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the Kite medical monitor
* Primary immunodeficiency
* History of autoimmune disease (eg, Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years prior to enrollment
* Known history of infection with human immunodeficiency virus (HIV), hepatitis B (HBsAg positive), or hepatitis C (anti-HCV positive). A history of treated hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative polymerase chain reaction (qPCR) and/or nucleic acid testing

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (9):
- United States (9):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kirtane K; Massarelli E; Hanna GJ; et al KITE-439: A Phase 1 Study of HPV16 E7 T Cell Receptor-engineered T Cells in Patients with Relapsed/Refractory HPV16-positive Cancers. ASCO Poster 2020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States.
Pre-assignment Details: 8 participants were screened. The study was terminated earlier than planned, and thus the study did not proceed to Phase 1B.
Groups:
- Phase 1A: 1 x 10^6 KITE-439 (Cohort 1): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, intravenous (IV) infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^6 E7 T-cell receptor (TCR) T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, subcutaneous (SC) injection, once on Days 0 to 6.
- Phase 1A: 3 x 10^6 KITE-439 (Cohort 2): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 3 × 10^6 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
- Phase 1A: 1 x 10^7 KITE-439 (Cohort 3): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^7 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
- Phase 1A: 3 x 10^7 KITE-439 (Cohort 4): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 3 × 10^7 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
- Phase 1A: 1 x 10^8 KITE-439 (Cohort 5): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^8 E7 TCR T cells/kg on Day 0 (maximum allowable dose was 5 × 10^9 E7 TCR T cells) along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
- Phase 1A: 1 x 10^8 KITE-439 (Cohort 6): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^8 E7 TCR T cells/kg on Day 0 (maximum allowable dose was 1 × 10^10 E7 TCR T cells) along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
Period: Overall Study
Arm/Group | Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) | Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) | Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) | Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 6)
Started | 1 | 1 | 1 | 1 | 3 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 3 | 1
Not completed — Death | 1 | 1 | 1 | 1 | 1 | 1
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Participant | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were treated with any dose of KITE-439.
Groups:
- Phase 1A: 1 x 10^6 KITE-439 (Cohort 1): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^6 E7 TCR T cells/kg on Day 0 along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
- Phase 1A: 1 x 10^8 KITE-439 (Cohort 6): Participants received conditioning chemotherapy of cyclophosphamide 30 mg/kg, IV infusion, once on Days -7 and -6 and fludarabine, 25 mg/m^2, IV infusion, once on Days -7 to -3 followed by KITE-439 infusion, up to 1 × 10^8 E7 TCR T cells/kg on Day 0 (maximum allowable dose was 1 ×10^10 E7 TCR T cells) along with the interleukin-2 of 2,50,000 IU/kg, SC injection, once on Days 0 to 6.
- Total: Total of all reporting groups
Arm/Group | Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) | Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) | Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) | Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 6) | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (NA) — Standard deviation cannot be calculated for single participant. | 54.0 (NA) — Standard deviation cannot be calculated for single participant. | 60.0 (NA) — Standard deviation cannot be calculated for single participant. | 77.0 (NA) — Standard deviation cannot be calculated for single participant. | 59.7 (9.45) | 40.0 (NA) — Standard deviation cannot be calculated for single participant. | 58.5 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Male | 1 | 1 | 1 | 1 | 1 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 3 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 1 | 3 | 1 | 8
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 1 | 1 | 3 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Phase 1A: Percentage of Participants Experiencing Adverse Events Defined as Dose-Limiting Toxicities (DLTs)
Description: A DLT is defined as protocol-defined KITE-439 related Grade 3 events with onset within the first 21 days following KITE-439 infusion and which do not resolve to ≤Grade 2 events within 48 hours, ≥Grade 4 events with onset within the first 21 days following KITE-439 infusion, regardless of duration.
Time Frame: First infusion date of KITE-439 up to 21 days
Population: DLT evaluable set included participants treated in Phase 1A who received the target dose (± 20%) and had the opportunity to be followed for at least 21 days after the KITE-439 infusion or received a dose of KITE-439 lower than the target dose and experienced a DLT within 21 days after the KITE-439 infusion.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) | Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) | Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) | Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 6)
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 1
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1B: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) as evaluated by modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Up to 1.4 years
Population: Due to early termination of study, Phase 1B dose of KITE-439 was not established and Phase 1B of study was not conducted.
Groups:
- Phase 1B: KITE-439: Participants were to receive cyclophosphamide and fludarabine conditioning chemotherapy followed by the investigational treatment, KITE-439, at a dose selected based on Phase 1A but the study was terminated before proceeding to Phase 1B.
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

3. Secondary Outcome: Phase 1B: Duration of Response (DOR)
Description: For participants who experience an objective response, DOR was defined as the time from the date of their first objective response to the date of disease progression per modified RECIST v1.1 or death from any cause.
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1B: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the KITE-439 infusion date to the date of disease progression per modified RECIST v1.1 or death from any cause.
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 1B: Overall Survival
Description: Overall survival was defined as the time from KITE-439 infusion to the date of death.
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 1B: Percentage of Participants Experiencing Adverse Events
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1B: Percentage of Participants With Anti-KITE-439 Antibodies
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 1B: Percentage of Participants With Replication-competent Retrovirus (RCR)
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 1B: Levels of E7 TCR T Cells
Time Frame: Up to 1.4 years
Population: as for outcome 2
Arm/Group | Phase 1B: KITE-439
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to last follow-up visit date of 18 February 2022 (maximum 1.4 years); Adverse Events: First infusion date of KITE-439 up to data cut-off date of 14 February 2022 (maximum 1.4 years).
Description: Safety analysis set included all participants who were treated with any dose of KITE-439.
Arm/Group | Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) | Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) | Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) | Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 6)
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 3/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 1/1 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) (N=1) | Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) (N=1) | Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) (N=1) | Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) (N=1) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) (N=3) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 6) (N=1)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1A: 1 x 10^6 KITE-439 (Cohort 1) (N=1) | Phase 1A: 3 x 10^6 KITE-439 (Cohort 2) (N=1) | Phase 1A: 1 x 10^7 KITE-439 (Cohort 3) (N=1) | Phase 1A: 3 x 10^7 KITE-439 (Cohort 4) (N=1) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 5) (N=3) | Phase 1A: 1 x 10^8 KITE-439 (Cohort 6) (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 2 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 1 | 2 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT03912831/Prot_SAP_000.pdf